CLINICAL TRIAL: NCT00335153
Title: An Open-Label, 12-Month Safety and Efficacy Study of Levodopa - Carbidopa Intestinal Gel in Levodopa-Responsive Subjects With Advanced Parkinson's Disease and Severe Motor Fluctuations Despite Optimized Treatment With Available Parkinson's Disease Medications
Brief Title: Levodopa-Carbidopa Intestinal Gel Open-Label Study in Advanced Parkinson's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Collaborators: Quintiles, Inc. (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S187.3.004; 2006-005186-18 (EudraCT Number)
Record Dates: First submitted 2006-06-08; First posted 2006-06-09 (Estimated); Results first posted 2015-01-16 (Estimated); Last update posted 2015-01-16 (Estimated); Status verified 2015-01

CONDITIONS: Advanced Parkinson's Disease
Keywords: severe motor fluctuations; levodopa; levodopa/carbidopa intestinal gel; efficacy; dyskinesia; Parkinson's Disease; carbidopa; DUOPA
MeSH Terms: conditions — Dyskinesias; Parkinson Disease | interventions — Jejunostomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Levodopa-Carbidopa Intestinal Gel (LCIG) (Experimental): All participants were to receive LCIG, via the NJ tube during the nasojejunal (NJ) Test Period and delivered to the proximal small intestine via percutaneous endoscopic gastrostomy - with jejunal extension tube (PEG-J) during the Post-PEG-J Long-Term Treatment Period. The starting dose was individually determined based on the daily dose of oral levodopa prior to study enrollment.
  The infusion dose was individually optimized for each participant on the basis of response and potential adverse events. During the Post-PEG-J Long-Term Treatment Period, LCIG was expected to be infused continuously over approximately 16 hours daily with a rate of infusion ranging from 1 to 10 mL/hour (20 to 200 mg of levodopa/hour), in most instances.
  Interventions: Drug: Levodopa-carbidopa intestinal gel; Device: CADD-Legacy® 1400 ambulatory infusion pump; Device: PEG tube; Device: J-tube

INTERVENTIONS:
Drug: Levodopa-carbidopa intestinal gel — Infusion should be kept within a range of 0.5-10 mL/hour (10-200 mg levodopa/hour) and is usually 2-6 mL/hour (40-120 mg levodopa/hour).
Device: CADD-Legacy® 1400 ambulatory infusion pump
Device: PEG tube — percutaneous endoscopic gastrostomy tube
Device: J-tube — jejunal tube

SUMMARY:
The primary objective of this study will be to provide further evidence of the long-term safety and tolerability of levodopa-carbidopa intestinal gel (Duodopa®) over 12-months in participants with advanced Parkinson's disease (PD) and severe motor fluctuations.

DETAILED DESCRIPTION:
The study was composed of a screening period followed by 3 sequential on-treatment periods, as follows:

* Screening Period (up to 28 days): determination of eligibility and discontinuation of antiparkinsonian disease medications other than levodopa-carbidopa immediate release (LC-oral) prior to nasojejunal (NJ) tube placement.
* NJ Test Period (2 to 14 days): first hospitalization period, Baseline assessments, placement of NJ tube, and optimization of levodopa-carbidopa intestinal gel (LCIG) treatment via NJ tube and infusion pump (participant was hospitalized for NJ tube placement but hospitalization was not required for entire duration of LCIG treatment optimization).
* PEG-J Period (2 to 14 days): second hospitalization period; placement of PEG-J tube; further optimization of LCIG treatment.
* Post PEG-J Long-Term Treatment Period (Day 28 to Day 378): LCIG administration via a permanent PEG-J tube and infusion pump, with dosage adjusted according to clinical condition.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic Parkinson's disease (PD) according to United Kingdom Parkinson's Disease Society (UKPDS) Brain Bank Criteria
* Levodopa-responsive with severe motor fluctuations
* Recognizable off and on state (motor fluctuations) confirmed by diary

Exclusion Criteria:

* Diagnosis is unclear or a suspicion of other parkinsonian syndromes exists such as secondary parkinsonism
* Undergone surgery for the treatment of PD
* Contraindications to levodopa (such as narrow angle glaucoma)

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 354 (Actual)
Dates: Start 2008-01; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janet Benesh, Study Director — AbbVie
Locations (83):
- United States (31):
  - Site Reference ID/Investigator# 50065, Birmingham, Alabama
  - Site Reference ID/Investigator# 50059, Fountain Valley, California
  - Site Reference ID/Investigator# 50048, Los Angeles, California
  - Site Reference ID/Investigator# 50076, Oceanside, California
  - Site Reference ID/Investigator# 50061, Englewood, Colorado
  - Site Reference ID/Investigator# 50079, Washington D.C., District of Columbia
  - Site Reference ID/Investigator# 50077, Bradenton, Florida
  - Site Reference ID/Investigator# 50060, Fort Lauderdale, Florida
  - Site Reference ID/Investigator# 50049, Gainesville, Florida
  - Site Reference ID/Investigator# 50047, Jacksonville, Florida
  - Site Reference ID/Investigator# 50068, Port Charlotte, Florida
  - Site Reference ID/Investigator# 50046, Tampa, Florida
  - Site Reference ID/Investigator# 50062, Augusta, Georgia
  - Site Reference ID/Investigator# 50050, Chicago, Illinois
  - Site Reference ID/Investigator# 50078, Chicago, Illinois
  - Site Reference ID/Investigator# 50064, Lexington, Kentucky
  - Site Reference ID/Investigator# 50075, Shreveport, Louisiana
  - Site Reference ID/Investigator# 50080, Baltimore, Maryland
  - Site Reference ID/Investigator# 50074, Baltimore, Maryland
  - Site Reference ID/Investigator# 50073, St Louis, Missouri
  - Site Reference ID/Investigator# 50042, Omaha, Nebraska
  - Site Reference ID/Investigator# 50072, Manhasset, New York
  - Site Reference ID/Investigator# 50067, New York, New York
  - Site Reference ID/Investigator# 50066, New York, New York
  - Site Reference ID/Investigator# 50069, Raleigh, North Carolina
  - Site Reference ID/Investigator# 50063, Winston-Salem, North Carolina
  - Site Reference ID/Investigator# 50043, Cincinnati, Ohio
  - Site Reference ID/Investigator# 50044, Cleveland, Ohio
  - Site Reference ID/Investigator# 50058, Burlington, Vermont
  - Site Reference ID/Investigator# 50045, Kirkland, Washington
  - Site Reference ID/Investigator# 50070, Milwaukee, Wisconsin
- Australia (3):
  - Site Reference ID/Investigator# 46429, Adelaide
  - Site Reference ID/Investigator# 46427, Heidelberg
  - Site Reference ID/Investigator# 46425, Westmead
- Canada (3):
  - Site Reference ID/Investigator# 54545, Edmonton
  - Site Reference ID/Investigator# 46433, Montreal
  - Site Reference ID/Investigator# 46434, Toronto
- Czechia (5):
  - Site Reference ID/Investigator# 46436, Brno
  - Site Reference ID/Investigator# 46438, Hradec Králové
  - Site Reference ID/Investigator# 46435, Pardubice
  - Site Reference ID/Investigator# 46437, Prague
  - Site Reference ID/Investigator# 46439, Prague
- Site Reference ID/Investigator# 48003, Lahti, Finland
- Germany (7):
  - Site Reference ID/Investigator# 48028, Berlin
  - Site Reference ID/Investigator# 48029, Berlin
  - Site Reference ID/Investigator# 48036, Freiburg im Breisgau
  - Site Reference ID/Investigator# 48034, Göttingen
  - Site Reference ID/Investigator# 48022, Hanau
  - Site Reference ID/Investigator# 48024, Hanover
  - Site Reference ID/Investigator# 48035, Mainz
- Site Reference ID/Investigator# 49882, Tel Aviv, Israel
- Italy (6):
  - Site Reference ID/Investigator# 50131, Arcugnano
  - Site Reference ID/Investigator# 50132, Catania
  - Site Reference ID/Investigator# 50128, Genoa
  - Site Reference ID/Investigator# 50129, Lido di Camaiore
  - Site Reference ID/Investigator# 50130, Naples
  - Site Reference ID/Investigator# 50127, Rome
- Site Reference ID/Investigator# 50138, Nijmegen, Netherlands
- New Zealand (4):
  - Site Reference ID/Investigator# 50126, Auckland
  - Site Reference ID/Investigator# 50123, Christchurch
  - Site Reference ID/Investigator# 50124, Hamilton
  - Site Reference ID/Investigator# 50125, Wellington
- Poland (2):
  - Site Reference ID/Investigator# 50140, Lodz
  - Site Reference ID/Investigator# 50139, Poznan
- Portugal (4):
  - Site Reference ID/Investigator# 50136, Almada
  - Site Reference ID/Investigator# 50134, Coimbra
  - Site Reference ID/Investigator# 50135, Lisbon
  - Site Reference ID/Investigator# 50137, Porto
- Russia (6):
  - Site Reference ID/Investigator# 50143, Kazan'
  - Site Reference ID/Investigator# 50141, Moscow
  - Site Reference ID/Investigator# 50145, Saint Petersburg
  - Site Reference ID/Investigator# 50142, Saint Petersburg
  - Site Reference ID/Investigator# 50147, Saint Petersburg
  - Site Reference ID/Investigator# 50146, Saint Petersburg
- Spain (5):
  - Site Reference ID/Investigator# 50154, Barcelona
  - Site Reference ID/Investigator# 50152, Barcelona
  - Site Reference ID/Investigator# 50202, Barcelona
  - Site Reference ID/Investigator# 50155, Barcelona
  - Site Reference ID/Investigator# 50153, Madrid
- Thailand (2):
  - Site Reference ID/Investigator# 50150, Bangkok
  - Site Reference ID/Investigator# 50151, Bangkok
- United Kingdom (2):
  - Site Reference ID/Investigator# 50149, Liverpool
  - Site Reference ID/Investigator# 50148, London

REFERENCES:
- [Derived] Chang FC, Kwan V, van der Poorten D, Mahant N, Wolfe N, Ha AD, Griffith JM, Tsui D, Kim SD, Fung VS. Intraduodenal levodopa-carbidopa intestinal gel infusion improves both motor performance and quality of life in advanced Parkinson's disease. J Clin Neurosci. 2016 Mar;25:41-5. doi: 10.1016/j.jocn.2015.05.059. Epub 2016 Jan 14. PMID 26777085
- [Derived] Lew MF, Slevin JT, Kruger R, Martinez Castrillo JC, Chatamra K, Dubow JS, Robieson WZ, Benesh JA, Fung VS. Initiation and dose optimization for levodopa-carbidopa intestinal gel: Insights from phase 3 clinical trials. Parkinsonism Relat Disord. 2015 Jul;21(7):742-8. doi: 10.1016/j.parkreldis.2015.04.022. Epub 2015 Apr 28. PMID 25962554
- [Derived] Fernandez HH, Standaert DG, Hauser RA, Lang AE, Fung VS, Klostermann F, Lew MF, Odin P, Steiger M, Yakupov EZ, Chouinard S, Suchowersky O, Dubow J, Hall CM, Chatamra K, Robieson WZ, Benesh JA, Espay AJ. Levodopa-carbidopa intestinal gel in advanced Parkinson's disease: final 12-month, open-label results. Mov Disord. 2015 Apr;30(4):500-9. doi: 10.1002/mds.26123. Epub 2014 Dec 24. PMID 25545465
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Levodopa-Carbidopa Intestinal Gel (LCIG): All participants were to receive levodopa-carbidopa intestinal gel (LCIG), via the nasojejunal (NJ) tube during the NJ Test Period and delivered to the proximal small intestine via percutaneous endoscopic gastrostomy with jejunal extension tube (PEG-J) during the Post-PEG-J Long-Term Treatment Period. The starting dose was individually determined based on the daily dose of oral levodopa prior to study enrollment.
  The infusion dose was individually optimized for each participant on the basis of response and potential adverse events. During the Post-PEG-J Long-Term Treatment Period, LCIG was expected to be infused continuously over approximately 16 hours daily with a rate of infusion ranging from 1 to 10 mL/hour (20 to 200 mg of levodopa/hour), in most instances.
Period: Nasojejunal (NJ) Test Period
Arm/Group | Levodopa-Carbidopa Intestinal Gel (LCIG)
Started | 354
Completed | 324
Not Completed | 30
Not completed — Adverse Event | 5
Not completed — Lack of Efficacy | 5
Not completed — Withdrawal by Subject | 12
Not completed — Administrative | 1
Not completed — Protocol Violation | 7
Period: Post-PEG-J Long-Term Treatment Period
Arm/Group | Levodopa-Carbidopa Intestinal Gel (LCIG)
Started | 324
Completed | 272
Not Completed | 52
Not completed — Adverse Event | 22
Not completed — Lack of Efficacy | 2
Not completed — Withdrawal by Subject | 13
Not completed — Administrative | 13
Not completed — Protocol Violation | 2

BASELINE CHARACTERISTICS:
Groups:
- Levodopa-Carbidopa Intestinal Gel (LCIG): All participants were to receive LCIG, via the NJ tube during the NJ Test Period and delivered to the proximal small intestine via PEG-J during the Post-PEG-J Long-Term Treatment Period. The starting dose was individually determined based on the daily dose of oral levodopa prior to study enrollment.
  The infusion dose was individually optimized for each participant on the basis of response and potential adverse events. During the Post-PEG-J Long-Term Treatment Period, LCIG was expected to be infused continuously over approximately 16 hours daily with a rate of infusion ranging from 1 to 10 mL/hour (20 to 200 mg of levodopa/hour), in most instances.
Arm/Group | Levodopa-Carbidopa Intestinal Gel (LCIG)
Number analyzed (Participants) | 354
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.1 (9.1)
Age, Customized [Number; unit: participants]
  <65 years | 171
  >=65 years | 183
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 152
  Male | 202

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs), Deaths and Discontinuations Due to AEs
Description: AE=any untoward medical occurrence which does not necessarily have a causal relationship with this treatment. SAE=any untoward medical occurrence that: results in death; is life-threatening (an event in which the subject was at risk of death at the time of the event); requires inpatient hospitalization or prolongation of an existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect; or other important medical events. Treatment-emergent events (TEAE or TESAE)=those starting after the first dose of study drug. Severe=severity reported as 'severe' or missing. Possibly or Probably Treatment Related=drug-event relationship reported as 'possible', 'probable' or missing. Death=a fatal outcome of an SAE or AE.
Time Frame: Screening through Day 378 + 30 days
Population: Safety Data Set: participants who were allocated to treatment, had started placement of NJ tube, and had at least 1 post-baseline safety evaluation (only participants lost to follow-up with no post-baseline information were excluded).
Measure: Number; unit: participants
Arm/Group | Levodopa-Carbidopa Intestinal Gel (LCIG)
Number analyzed (Participants) | 354
participants
  Deaths | 8
  TE Deaths | 7
  >=1 SAE | 111
  >=1TESAE | 108
  >=1 TEAE Leading to Study Termination | 27
  >=1 TEAE | 323
  >=1 Severe TEAE | 102
  >=1 Possibly or Probably Treatment Related TEAE | 272
  No TEAE | 31

2. Primary Outcome: Number of Participants With Device Complications During the Nasojejunal (NJ) Test Period
Description: Complications of the infusion device were collected during the NJ Test period. Pump, intestinal tube, NJ tube, and other complications included (but were not limited to) device breakage, device leakage, device malfunction, device misuse, device occlusion, intentional and unintentional device removal by participant, complication of device insertion, device dislocation, device breakage, device dislocation, and post-procedural hemorrhage.
Time Frame: NJ Test Period (from 2 to 14 days)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Levodopa-Carbidopa Intestinal Gel (LCIG)
Number analyzed (Participants) | 354
participants
  >=1 Complication | 90
  Pump Complication | 7
  Intestinal Tube Complication | 4
  NJ Tube Complication | 68
  Other Complications | 25

3. Primary Outcome: Number of Participants With Device Complications During the Percutaneous Endoscopic Gastrostomy - With Jejunal Extension Tube (PEG-J) Surgery and Post-PEG Long Term Treatment Periods
Description: Complications of the infusion device were collected during the PEG-J Surgery and Post-PEG Long-Term Treatment periods. Pump, PEG-J, stoma, and other complications included (but were not limited to) device breakage, device leakage, device malfunction, device misuse, device occlusion, intentional and unintentional device removal by participant, complication of device insertion, device dislocation, device breakage, device dislocation, and post-procedural hemorrhage.
Time Frame: PEG-J Surgery Period (from 2 to 14 days) through the Long Term Treatment Period (Day 28 to Day 378)
Population: Post-PEG Safety Data Set: participants who continued to the PEG-J surgery, and had at least 1 post-baseline safety evaluation (only participants lost to follow-up with no post-baseline information were excluded).
Measure: Number; unit: participants
Arm/Group | Levodopa-Carbidopa Intestinal Gel (LCIG)
Number analyzed (Participants) | 324
participants
  >=1 Complication | 282
  Pump Complication | 116
  Intestinal Tube Complication | 165
  PEG-J Complication | 114
  Stoma Complication | 116
  Other Complication | 114

4. Primary Outcome: Number of Participants With Potentially Clinically Significant Values for Hematology Parameters
Description: Potentially clinically significant values for red blood cells (RBCs), hemoglobin, and hematocrit are specified for females (f) and males (m) separately in the category rows.
Time Frame: Screening through Day 378
Population: Post-PEG Safety Data Set: participants who continued to the PEG-J surgery, and had at least 1 post-baseline safety evaluation (only participants lost to follow-up with no post-baseline information were excluded); n=number of participants with assessment.
Measure: Number; unit: participants
Arm/Group | Levodopa-Carbidopa Intestinal Gel (LCIG)
Number analyzed (Participants) | 324
participants
  RBCs <2.0*10^12/L (f), <2.5*10^12/L (m); n=316 | 0
  Hemoglobin <90 g/L (f), <100 g/L (m); n=316 | 4
  Hematocrit <30% (f), <34% (m); n=315 | 27
  White Blood Cells <2.8*10^9/L; n=316 | 3
  White Blood Cells >16.0*10^9/L; n=316 | 0
  Neutrophils <1.2*10^9/L; n=316 | 0
  Lymphocytes <0.75*10^9/L; n=316 | 21
  Lymphocytes >80%; n=316 | 0
  Platelet Count <95*10^9/L; n=315 | 1
  Platelet Count >700*10^9/L; n=315 | 0
  Mean Corpuscular Volume <60 fL; n=315 | 0
  Mean Corpuscular Volume >120 fL; n=315 | 0
  Eosinophils >10%; n=316 | 7
  Monocytes >30%; n=316 | 0

5. Primary Outcome: Number of Participants With Potentially Clinically Significant Values for Clinical Chemistry Parameters
Description: Terms abbreviated in the table include aspartate aminotransferase (AST), upper limit of normal (ULN), alanine aminotransferase (ALT), gamma-glutamyl transpeptidase (GGT), lactate dehydrogenase (LDH), blood urea nitrogen (BUN), female (f), and male (m).
Time Frame: Screening through Day 378
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Levodopa-Carbidopa Intestinal Gel (LCIG)
Number analyzed (Participants) | 324
participants
  AST >3*ULN; n=315 | 1
  ALT >3*ULN; n=315 | 0
  GGT >3*ULN; n=315 | 3
  LDH >3*ULN; n=315 | 0
  Alkaline Phosphatase >400 U/L; n=315 | 0
  Total Protein <45 g/L; n=315 | 0
  Total Bilirubin >2*ULN; n=315 | 0
  Creatine Kinase >3*ULN; n=315 | 7
  Sodium <126 mmol/L; n=315 | 2
  Sodium >156 mmol/L; n=315 | 2
  Potassium <3.0 mmol/L; n=315 | 1
  Potassium >6.0 mmol/L; n=315 | 1
  Calcium <1.75 mmol/L; n=315 | 2
  Calcium >3.0 mmol/L; n=315 | 0
  BUN >10.8 mmol/L; n=77 | 4
  Creatinine >177 mcmol/L; n=315 | 3
  Uric Acid >500 mcmol/L (f), >590 mcmol/L (m);n=315 | 0
  Glucose (nonfasting) <2.78 mmol/L; n=315 | 1
  Glucose (nonfasting) >16.0 mmol/L; n=315 | 1
  Cholesterol >12.9 mmol/L; n=315 | 0
  Triglycerides >5.6 mmol/L; n=315 | 2

6. Primary Outcome: Number of Participants With Potentially Clinically Significant Vital Sign Parameters
Description: Terms abbreviated in the table include supine systolic blood pressure (SuSBP), standing systolic blood pressure (StSBP), orthostatic systolic blood pressure (OSBP), supine diastolic blood pressure (SuDBP), standing diastolic blood pressure (StDBP), orthostatic diastolic blood pressure (ODBP), supine pulse (SuP) in beats per minute (bpm), standing pulse (StP), and body temperature (Temp). Increase and decrease are signified by ↑ and ↓, respectively.
Time Frame: up to 56 weeks
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Levodopa-Carbidopa Intestinal Gel (LCIG)
Number analyzed (Participants) | 324
participants
  SuSBP >=180 and >40 mm Hg ↑ from BL; n=324 | 4
  SuSBP <=90 and >30 mm Hg ↓ from BL; n=324 | 17
  StSBP >=180 and >40 mm Hg ↑ from BL; n=324 | 2
  StSBP <=90 and >30 mm Hg ↓ from BL; n=324 | 35
  OSBP: ↓ >=30 mm Hg (Supine to Standing); n=324 | 80
  SuDBP >=105 and >30 mm Hg ↑ from BL; n=324 | 5
  SuDBP <=50 and >30 mm Hg ↓ from BL; n=324 | 11
  StDBP >=105 and >30 mm Hg ↑ from BL; n=324 | 8
  StDBP <=50 and >30 mm Hg ↓ from BL; n=324 | 12
  ODBP: ↓ >=20 mm Hg (Supine to Standing); n=324 | 59
  SuP >=120 and >30 bpm ↑ from BL; n=324 | 0
  SuP <=50 and >30 bpm ↓ from BL; n=324 | 1
  StP >=120 and >30 bpm ↑ from BL; n=324 | 0
  StP <=50 and >30 bpm ↓ from BL; n=324 | 0
  Temp >=38.3 and >1.1°C ↑ from BL; n=322 | 2
  Weight >=7% ↑ from BL; n=272 | 25
  Weight <=7% ↓ from BL; n=272 | 79

7. Primary Outcome: Number of Participants With Potentially Clinically Significant Electrocardiogram (ECG) Parameters
Description: Terms abbreviated in the table include heart rate (HR) in beats per minute (bpm), PR interval (PRI), QT interval corrected for heart rate using Bazett's formula (QTcB), and QT interval corrected for heart rate using Fridericia's formula (QTcF). Increase and decrease are signified by ↑ and ↓, respectively.
Time Frame: Screening through Day 378
Population: Post-PEG Safety Data Set: participants who continued to the PEG-J surgery, and had at least 1 post-baseline safety evaluation (only participants lost to follow-up with no post-baseline information were excluded); n=number of participants with given assessment.
Measure: Number; unit: participants
Arm/Group | Levodopa-Carbidopa Intestinal Gel (LCIG)
Number analyzed (Participants) | 324
participants
  HR <=50 and >30 bpm ↓ from BL; n=321 | 1
  HR >=120 and >30 bpm ↑ from BL; n=321 | 1
  PR Interval <120 msec; n=321 | 6
  PR Interval >220 msec; n=321 | 26
  QTcB Interval >480 msec; n=319 | 15
  QTcB Interval >60 msec ↑ from BL; n=309 | 4
  QTcF Interval >480 msec; n=319 | 7
  QTcF Interval >60 msec ↑ from BL; n=309 | 3

8. Primary Outcome: Number of Participants With Sleep Attacks at Baseline
Description: To prospectively monitor for the possible development of sleep attacks, participants were asked if they had experienced any events in which they fell asleep suddenly or unexpectedly, including while engaged in some activity (e.g., eating/drinking, speaking, or driving) or at rest, with or without any previous warning of sleepiness. Those participants who reported 1 or more sleep attacks were asked to report the number of sleep attacks they experienced, whether they experienced sleepiness or drowsiness prior to the sleep attack, whether they experienced a 'bad' outcome or problem due to a sleep attack, and if so, how many 'bad' outcomes or problems they experienced.
Time Frame: Baseline
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Levodopa-Carbidopa Intestinal Gel (LCIG)
Number analyzed (Participants) | 324
participants
  Participants with >=1 Sleep Attacks | 7
  Number of Sleep Attacks Per Participant=1 | 4
  Number of Sleep Attacks Per Participant=2 | 0
  Number of Sleep Attacks Per Participant=3 | 0
  Number of Sleep Attacks Per Participant>3 | 2
  Number of Sleep Attacks Per Participant=Missing | 1
  Sleepiness/Drowsiness Prior to Sleep Attack | 4
  Bad Outcome/Problem Due to Sleep Attack | 1
  Number of Bad Outcomes/Problems=1 | 1
  Number of Bad Outcomes/Problems=2 | 0
  Number of Bad Outcomes/Problems=3 | 0
  Number of Bad Outcomes/Problems>3 | 0

9. Primary Outcome: Number of Participants With Sleep Attacks During the Post-PEG Long-Term Treatment Period
Description: as for outcome 8
Time Frame: During the Post-PEG Long-Term Treatment Period (Day 28 through Day 378)
Population: Post-PEG Safety Data Set: participants who continued to the PEG-J surgery, and had at least 1 post-baseline safety evaluation (only participants lost to follow-up with no post-baseline information were excluded) who had an assessment.
Measure: Number; unit: participants
Arm/Group | Levodopa-Carbidopa Intestinal Gel (LCIG)
Number analyzed (Participants) | 321
participants
  Participants with >=1 Sleep Attacks | 27
  Number of Sleep Attacks Per Participant=1 | 11
  Number of Sleep Attacks Per Participant=2 | 2
  Number of Sleep Attacks Per Participant=3 | 5
  Number of Sleep Attacks Per Participant>3 | 9
  Sleepiness/Drowsiness Prior to Sleep Attack | 11
  Bad Outcome/Problem Due to Sleep Attack | 2
  Number of Bad Outcomes/Problems=1 | 2
  Number of Bad Outcomes/Problems=2 | 0
  Number of Bad Outcomes/Problems=3 | 0
  Number of Bad Outcomes/Problems>3 | 0

10. Primary Outcome: Summary of Minnesota Impulsive Disorder Interview (MIDI) Assessment of Intense Impulsive Behavior at Baseline (BL) and During the Post-PEG Long-term Treatment (PPLT) Period
Description: The MIDI is a validated assessment of impulsive behavior consisting of a semistructured clinical interview assessing pathological gambling, trichotillomania (compulsive hair-pulling), kleptomania (compulsive stealing), pyromania (compulsive fire setting), intermittent explosive disorder, compulsive buying, and compulsive sexual behavior.
Time Frame: Baseline, during the Post-PEG Long-term Treatment Period (Day 28 through Day 378)
Population: Post-PEG Safety Data Set: participants who continued to the PEG-J surgery, and had at least 1 post-baseline safety evaluation (only participants lost to follow-up with no post-baseline information were excluded); n=number of participants with an assessment at timepoint.
Measure: Number; unit: participants
Arm/Group | Levodopa-Carbidopa Intestinal Gel (LCIG)
Number analyzed (Participants) | 324
participants
  BL Compulsive Buying; n=322 | 0
  BL Kleptomania; n=322 | 0
  BL Trichotillomania; n=322 | 0
  BL Intermittent Explosive Disorder; n=322 | 0
  BL Pyromania; n=322 | 0
  BL Pathological Gambling; n=322 | 2
  BL Compulsive Sexual Behavior; n=322 | 9
  PPLT Compulsive Buying; n=318 | 3
  PPLT Kleptomania; n=318 | 0
  PPLT Trichotillomania; n=318 | 0
  PPLT Intermittent Explosive Disorder; n=318 | 0
  PPLT Pyromania; n=318 | 0
  PPLT Pathological Gambling; n=318 | 6
  PPLT Compulsive Sexual Behavior; n=318 | 11

11. Primary Outcome: Change From Baseline in Abnormal Involuntary Movement Scale (AIMS) Total Score at Endpoint
Description: The AIMS is an investigator-completed rating scale that has a total of 12 items rating involuntary movements of various areas of the participant's body. Items 1 through 10 are rated on a 5-point scale of severity from 0 (none), 1 (minimal), 2 (mild), 3 (moderate), to 4 (severe), and items 11 and 12 are yes/no questions regarding issues with teeth or dentures. The total AIMS score was calculated by summing items 1-10, with a possible range of 0-40; a negative change indicates improvement. The AIMS was to be performed at consistent times, when the subject was experiencing his/her worst "On" time (dyskinesia [involuntary muscle movement]).
Time Frame: Baseline, Endpoint (last Post-PEG Long-Term Period visit up to Day 378)
Population: Post-PEG Safety Data Set: participants who continued to the PEG-J surgery, and had at least 1 post-baseline safety evaluation (only participants lost to follow-up with no post-baseline information were excluded); n=number of participants with assessment at timepoint.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Levodopa-Carbidopa Intestinal Gel (LCIG)
Number analyzed (Participants) | 324
units on a scale
  Baseline; n=318 | 9.6 (8.1)
  Change from Baseline at Endpoint; n=317 | -1.7 (9.0)

12. Secondary Outcome: Change From Baseline in Average Daily "Off" Time at Endpoint
Description: Based on the Parkinson's Disease Symptom Diary. "On" time is when PD symptoms are well controlled by the drug. "Off" time is when PD symptoms are not adequately controlled by the drug. The diary is completed every 30 minutes for the full 24 hours of each of 3 days prior to selected clinic visits. It reflects both time awake and time asleep. Daily totals are normalized to a 16-hour scale (i.e. 16 hours of awake time). The normalized totals for the 3 days prior to the visit are averaged for the analysis. Negative change from baseline for "off" time indicates improvement.
Time Frame: Baseline, Endpoint (last post-baseline visit up to Day 378)
Population: Full Analysis Data Set: participants who had at least 1 post-baseline safety evaluation, a baseline efficacy evaluation, and had data for at least 1 post-baseline assessment of this efficacy measurement during the Post-PEG Long-Term Treatment Period.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Levodopa-Carbidopa Intestinal Gel (LCIG)
Number analyzed (Participants) | 307
hours
  Baseline | 6.77 (2.37)
  Change from Baseline at Endpoint | -4.44 (2.89)
Statistical Analysis 1: Comparison: Levodopa-Carbidopa Intestinal Gel (LCIG); Test type: Superiority or Other; p < 0.001, t-test, 2 sided

13. Secondary Outcome: Change From Baseline in Average Daily Normalized "On" Time With Troublesome Dyskinesia at Endpoint
Description: Based on the Parkinson's Disease Symptom Diary. "On" time is when PD symptoms are well controlled by the drug. "Off" time is when PD symptoms are not adequately controlled by the drug. The diary is completed every 30 minutes for the full 24 hours of each of 3 days prior to selected clinic visits. It reflects both time awake and time asleep. Daily totals are normalized to a 16-hour scale (i.e. 16 hours of awake time). The normalized totals for the 3 days prior to the visit are averaged for the analysis.
Time Frame: Baseline, Endpoint (last post-baseline visit up to Day 378)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Levodopa-Carbidopa Intestinal Gel (LCIG)
Number analyzed (Participants) | 307
hours
  Baseline | 1.60 (2.03)
  Change from Baseline at Endpoint | -0.36 (2.77)
Statistical Analysis 1: Comparison: Levodopa-Carbidopa Intestinal Gel (LCIG); Test type: Superiority or Other; p = 0.023, t-test, 2 sided

14. Secondary Outcome: Change From Baseline in Average Daily "On" Time Without Troublesome Dyskinesia at Endpoint
Description: Based on the Parkinson's Disease Symptom Diary. "On" time is when PD symptoms are well controlled by the drug. "Off" time is when PD symptoms are not adequately controlled by the drug. "On" time without troublesome dyskinesia (involuntary muscle movement) is defined as "on" time without dyskinesia and "on" time with non-troublesome dyskinesia. The diary is completed every 30 minutes for the full 24 hours of each of 3 days prior to selected clinic visits. It reflects both time awake and time asleep. Daily totals are normalized to a 16-hour scale (i.e. 16 hours of awake time). The normalized totals for the 3 days prior to the visit are averaged for the analysis. Positive change from Baseline for "on" time without troublesome dyskinesia indicates improvement.
Time Frame: Baseline, Endpoint (last post-baseline visit up to Day 378)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Levodopa-Carbidopa Intestinal Gel (LCIG)
Number analyzed (Participants) | 307
hours
  Baseline | 4.83 (2.72)
  Change from Baseline at Endpoint | 3.86 (4.65)
Statistical Analysis 1: Comparison: Levodopa-Carbidopa Intestinal Gel (LCIG); Test type: Superiority or Other; p < 0.001, t-test, 2 sided

15. Secondary Outcome: Clinical Global Impression - Status (CGI-S) Score at Baseline and Clinical Global Impression - Improvement (CGI-I) Score at Endpoint
Description: The CGI-S is a global assessment by the Investigator of current symptomatology and impact of illness on functioning. The ratings of the CGI-S are as follows: 1 = normal, 2 = borderline ill, 3 = mildly ill, 4 = moderately ill, 5 = markedly ill, 6 = severely ill, and 7 = among the most extremely ill. The CGI-I is a global assessment by the Investigator of the change in clinical status since the start of treatment. The CGI-I ratings are as follows: 1 = very much improved, 2 = much improved, 3 = minimally improved, 4 = no change, 5 = minimally worse, 6 = much worse, 7 = very much worse.
Time Frame: Baseline, Endpoint (last post-baseline visit up to Day 378)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Levodopa-Carbidopa Intestinal Gel (LCIG)
Number analyzed (Participants) | 316
units on a scale
  CGI-S Baseline | 4.85 (0.84)
  CGI-I at Endpoint | 2.10 (0.95)
Statistical Analysis 1: Comparison: Levodopa-Carbidopa Intestinal Gel (LCIG); Test type: Superiority or Other; p < 0.001, t-test, 2 sided

16. Secondary Outcome: Change From Baseline in Unified Parkinson's Disease Rating Scale (UPDRS) Part I Score at Month 12
Description: The UPDRS is an Investigator-used rating tool to follow the longitudinal course of Parkinson's disease. The Part I Score is the sum of the answers to the 4 questions that comprise Part I, each of which are measured on a 5-point scale (0-4). The Part I score ranges from 0-16 and higher scores are associated with more disability.
Time Frame: Baseline, Endpoint (last post-baseline visit up to Day 378)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Levodopa-Carbidopa Intestinal Gel (LCIG)
Number analyzed (Participants) | 288
units on a scale
  Baseline | 2.2 (1.9)
  Change from Baseline at Endpoint | 0.0 (1.8)
Statistical Analysis 1: Comparison: Levodopa-Carbidopa Intestinal Gel (LCIG); Test type: Superiority or Other; p = 0.974, t-test, 2 sided

17. Secondary Outcome: Change From Baseline in Unified Parkinson's Disease Rating Scale (UPDRS) Part II Score at Endpoint
Description: The UPDRS is an Investigator-used rating tool to follow the longitudinal course of Parkinson's disease. The Part II score is the sum of the answers to the 13 questions that comprise Part II, each of which are measured on a 5-point scale (0-4). The Part II score ranges from 0-52 and higher scores are associated with more disability.
Time Frame: Baseline, Endpoint (last post-baseline visit up to Day 378)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Levodopa-Carbidopa Intestinal Gel (LCIG)
Number analyzed (Participants) | 288
units on a scale
  Baseline | 17.5 (6.7)
  Change from Baseline at Endpoint | -4.4 (6.5)
Statistical Analysis 1: Comparison: Levodopa-Carbidopa Intestinal Gel (LCIG); Test type: Superiority or Other; p < 0.001, t-test, 2 sided

18. Secondary Outcome: Change From Baseline in Unified Parkinson's Disease Rating Scale (UPDRS) Part III Score at Endpoint
Description: The UPDRS is an Investigator-used rating tool to follow the longitudinal course of Parkinson's disease. The Part III score is the sum of the 27 answers provided to the 14 Part III questions, each of which are measured on a 5-point scale (0-4). The Part III score ranges from 0-108 and higher scores are associated with more disability.
Time Frame: Baseline, Endpoint (last post-baseline visit up to Day 378)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Levodopa-Carbidopa Intestinal Gel (LCIG)
Number analyzed (Participants) | 286
units on a scale
  Baseline | 28.9 (13.7)
  Change from Baseline at Endpoint | -7.4 (13.2)
Statistical Analysis 1: Comparison: Levodopa-Carbidopa Intestinal Gel (LCIG); Test type: Superiority or Other; p < 0.001, t-test, 2 sided

19. Secondary Outcome: Change From Baseline in Unified Parkinson's Disease Rating Scale (UPDRS) Total Score at Endpoint
Description: The UPDRS is an Investigator-used rating tool to follow the longitudinal course of Parkinson's disease. The total score is the sum of the responses to the 31 questions (44 answers) that comprise Parts I-III of the scale. The total score will range from 0-176, with 176 representing the worst (total) disability, and 0 representing no disability.
Time Frame: Baseline, Endpoint (last post-baseline visit up to Day 378)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Levodopa-Carbidopa Intestinal Gel (LCIG)
Number analyzed (Participants) | 287
units on a scale
  Baseline | 48.6 (18.9)
  Change from Baseline at Endpoint | -11.7 (18.3)
Statistical Analysis 1: Comparison: Levodopa-Carbidopa Intestinal Gel (LCIG); Test type: Superiority or Other; p < 0.001, t-test, 2 sided

20. Secondary Outcome: Change From Baseline in Unified Parkinson's Disease Rating Scale (UPDRS) Part IV Score at Endpoint
Description: The UPDRS is an Investigator-used rating tool to follow the longitudinal course of Parkinson's disease. The Part IV Score is the sum of the answers to the 11 questions that comprise Part IV, each of which are measured on a 5-point scale (0-4) or a 2-point scale (0 or 1). The Part IV score ranges from 0-23 and higher scores are associated with more disability.
Time Frame: Baseline, Endpoint (last post-baseline visit up to Day 378)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Levodopa-Carbidopa Intestinal Gel (LCIG)
Number analyzed (Participants) | 287
units on a scale
  Baseline | 9.2 (2.9)
  Change from Baseline at Endpoint | -3.5 (3.5)
Statistical Analysis 1: Comparison: Levodopa-Carbidopa Intestinal Gel (LCIG); Test type: Superiority or Other; p < 0.001, t-test, 2 sided

21. Secondary Outcome: Change From Baseline in Parkinson's Disease Questionnaire (PDQ-39) Summary Index at Endpoint
Description: The PDQ-39 is a self-administered questionnaire which comprises 39 items addressing 8 domains of health in Parkinson's disease patients. These include: mobility, activities of daily living, emotional well-being, stigma, social support, cognition, communication, and bodily discomfort. The PDQ-39 Summary Index is the sum of all answers divided by the highest score possible (i.e. number of answers multiplied by 4) which is multiplied by 100 to put the score on a 0-100 scale. Higher scores are associated with more severe symptoms.
Time Frame: Baseline, Endpoint (last post-baseline visit up to Day 378)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Levodopa-Carbidopa Intestinal Gel (LCIG)
Number analyzed (Participants) | 317
units on a scale
  Baseline | 42.7 (15.0)
  Change from Baseline at Endpoint | -6.9 (14.1)
Statistical Analysis 1: Comparison: Levodopa-Carbidopa Intestinal Gel (LCIG); Test type: Superiority or Other; p < 0.001, t-test, 2 sided

22. Secondary Outcome: Change From Baseline in Parkinson's Disease Questionnaire (PDQ-39) Mobility Domain Score at Endpoint
Description: The PDQ-39 is a self-administered questionnaire which comprises 39 items addressing 8 domains of health in Parkinson's disease patients. The PDQ-39 Domain: Mobility (e.g., fear of falling when walking) includes 10 questions, each answered on a 5-point scale. The domain scores are calculated by first summing the answers to the questions in the domain. The sum is divided by the highest score possible (i.e., number of answers multiplied by 4) and the quotient is multiplied by 100 to put the score on a scale from 0 to 100, where lower scores indicate a better perceived health status. Higher scores are consistently associated with the more severe symptoms of the disease such as tremor and stiffness.
Time Frame: Baseline, Endpoint (last post-baseline visit up to Day 378)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Levodopa-Carbidopa Intestinal Gel (LCIG)
Number analyzed (Participants) | 317
units on a scale
  Baseline | 58.8 (22.8)
  Change from Baseline at Endpoint | -11.2 (23.4)
Statistical Analysis 1: Comparison: Levodopa-Carbidopa Intestinal Gel (LCIG); Test type: Superiority or Other; p < 0.001, t-test, 2 sided

23. Secondary Outcome: Change From Baseline in Parkinson's Disease Questionnaire (PDQ-39) Activities of Daily Living Domain Score at Endpoint
Description: The PDQ-39 is a self-administered questionnaire which comprises 39 items addressing 8 domains of health in Parkinson's disease patients. The PDQ-39 Domain: Activities of Daily Living (e.g., difficulty cutting food) includes 6 questions, each answered on a 5-point scale. The domain scores are calculated by first summing the answers to the questions in the domain. The sum is divided by the highest score possible (i.e., number of answers multiplied by 4) and the quotient is multiplied by 100 to put the score on a scale from 0 to 100, where lower scores indicate a better perceived health status. Higher scores are consistently associated with the more severe symptoms of the disease such as tremor and stiffness.
Time Frame: Baseline, Endpoint (last post-baseline visit up to Day 378)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Levodopa-Carbidopa Intestinal Gel (LCIG)
Number analyzed (Participants) | 317
units on a scale
  Baseline | 50.7 (22.3)
  Change from Baseline at Endpoint | -8.3 (22.6)
Statistical Analysis 1: Comparison: Levodopa-Carbidopa Intestinal Gel (LCIG); Test type: Superiority or Other; p < 0.001, t-test, 2 sided

24. Secondary Outcome: Change From Baseline in Parkinson's Disease Questionnaire (PDQ-39) Emotional Well-Being Domain Score at Endpoint
Description: The PDQ-39 is a self-administered questionnaire which comprises 39 items addressing 8 domains of health in Parkinson's disease patients. The PDQ-39 Domain: Emotional Well-being (e.g., feelings of isolation) includes 6 questions, each answered on a 5-point scale. The domain scores are calculated by first summing the answers to the questions in the domain. The sum is divided by the highest score possible (i.e., number of answers multiplied by 4) and the quotient is multiplied by 100 to put the score on a scale from 0 to 100, where lower scores indicate a better perceived health status. Higher scores are consistently associated with the more severe symptoms of the disease such as tremor and stiffness.
Time Frame: Baseline, Endpoint (last post-baseline visit up to Day 378)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Levodopa-Carbidopa Intestinal Gel (LCIG)
Number analyzed (Participants) | 317
units on a scale
  Baseline | 39.4 (21.8)
  Change from Baseline at Endpoint | -4.2 (19.7)
Statistical Analysis 1: Comparison: Levodopa-Carbidopa Intestinal Gel (LCIG); Test type: Superiority or Other; p < 0.001, t-test, 2 sided

25. Secondary Outcome: Change From Baseline in Parkinson's Disease Questionnaire (PDQ-39) Stigma Domain Score at Endpoint
Description: The PDQ-39 is a self-administered questionnaire which comprises 39 items addressing 8 domains of health in Parkinson's disease patients. The PDQ-39 Domain: Stigma (e.g., social embarrassment) consists of 4 questions, each answered on a 5-point scale. The domain scores are calculated by first summing the answers to the questions in the domain. The sum is divided by the highest score possible (i.e., number of answers multiplied by 4) and the quotient is multiplied by 100 to put the score on a scale from 0 to 100, where lower scores indicate a better perceived health status. Higher scores are consistently associated with the more severe symptoms of the disease such as tremor and stiffness.
Time Frame: Baseline, Endpoint (last post-baseline visit up to Day 378)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Levodopa-Carbidopa Intestinal Gel (LCIG)
Number analyzed (Participants) | 317
units on a scale
  Baseline | 32.5 (26.0)
  CHange from Baseline at Endpoint | -9.1 (22.1)
Statistical Analysis 1: Comparison: Levodopa-Carbidopa Intestinal Gel (LCIG); Test type: Superiority or Other; p < 0.001, t-test, 2 sided

26. Secondary Outcome: Change From Baseline in Parkinson's Disease Questionnaire (PDQ-39) Social Support Domain Score at Endpoint
Description: The PDQ-39 is a self-administered questionnaire which comprises 39 items addressing 8 domains of health in Parkinson's disease patients. The PDQ-39 Domain: Social Support includes 3 questions, each answered on a 5-point scale. The domain scores are calculated by first summing the answers to the questions in the domain. The sum is divided by the highest score possible (i.e., number of answers multiplied by 4) and the quotient is multiplied by 100 to put the score on a scale from 0 to 100, where lower scores indicate a better perceived health status. Higher scores are consistently associated with the more severe symptoms of the disease such as tremor and stiffness.
Time Frame: Baseline, Endpoint (last post-baseline visit up to Day 378)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Levodopa-Carbidopa Intestinal Gel (LCIG)
Number analyzed (Participants) | 315
units on a scale
  Baseline | 17.2 (19.7)
  Change from Baseline at Endpoint | -0.3 (18.9)
Statistical Analysis 1: Comparison: Levodopa-Carbidopa Intestinal Gel (LCIG); Test type: Superiority or Other; p = 0.757, t-test, 2 sided

27. Secondary Outcome: Change From Baseline in Parkinson's Disease Questionnaire (PDQ-39) Cognition Domain Score at Endpoint
Description: The PDQ-39 is a self-administered questionnaire which comprises 39 items addressing 8 domains of health in Parkinson's disease patients. The PDQ-39 Domain: Cognition includes 4 questions, each answered on a 5-point scale. The domain scores are calculated by first summing the answers to the questions in the domain. The sum is divided by the highest score possible (i.e., number of answers multiplied by 4) and the quotient is multiplied by 100 to put the score on a scale from 0 to 100, where lower scores indicate a better perceived health status. Higher scores are consistently associated with the more severe symptoms of the disease such as tremor and stiffness.
Time Frame: Baseline, Endpoint (last post-baseline visit up to Day 378)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Levodopa-Carbidopa Intestinal Gel (LCIG)
Number analyzed (Participants) | 317
units on a scale
  Baseline | 27.2 (18.6)
  Change from Baseline to Endpoint | -4.5 (18.0)
Statistical Analysis 1: Comparison: Levodopa-Carbidopa Intestinal Gel (LCIG); Test type: Superiority or Other; p < 0.001, t-test, 2 sided

28. Secondary Outcome: Change From Baseline in Parkinson's Disease Questionnaire (PDQ-39) Communication Domain Score at Endpoint
Description: The PDQ-39 is a self-administered questionnaire which comprises 39 items addressing 8 domains of health in Parkinson's disease patients. The PDQ-39 Domain: Communication includes 3 questions, each answered on a 5-point scale. The domain scores are calculated by first summing the answers to the questions in the domain. The sum is divided by the highest score possible (i.e., number of answers multiplied by 4) and the quotient is multiplied by 100 to put the score on a scale from 0 to 100, where lower scores indicate a better perceived health status. Higher scores are consistently associated with the more severe symptoms of the disease such as tremor and stiffness.
Time Frame: Baseline, Endpoint (last post-baseline visit up to Day 378)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Levodopa-Carbidopa Intestinal Gel (LCIG)
Number analyzed (Participants) | 317
units on a scale
  Baseline | 34.3 (20.4)
  Change from Baseline at Endpoint | -3.9 (19.4)
Statistical Analysis 1: Comparison: Levodopa-Carbidopa Intestinal Gel (LCIG); Test type: Superiority or Other; p < 0.001, t-test, 2 sided

29. Secondary Outcome: Change From Baseline in Parkinson's Disease Questionnaire (PDQ-39) Bodily Discomfort Domain Score at Endpoint
Description: The PDQ-39 is a self-administered questionnaire which comprises 39 items addressing 8 domains of health in Parkinson's disease patients. The PDQ-39 Domain: Bodily Discomfort includes 3 questions, each answered on a 5-point scale. The domain scores are calculated by first summing the answers to the questions in the domain. The sum is divided by the highest score possible (i.e., number of answers multiplied by 4) and the quotient is multiplied by 100 to put the score on a scale from 0 to 100, where lower scores indicate a better perceived health status. Higher scores are consistently associated with the more severe symptoms of the disease such as tremor and stiffness.
Time Frame: Baseline, Endpoint (last post-baseline visit up to Day 378)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Levodopa-Carbidopa Intestinal Gel (LCIG)
Number analyzed (Participants) | 317
units on a scale
  Baseline | 46.2 (22.9)
  Change from Baseline at Endpoint | -5.8 (22.4)
Statistical Analysis 1: Comparison: Levodopa-Carbidopa Intestinal Gel (LCIG); Test type: Superiority or Other; p < 0.001, t-test, 2 sided

30. Secondary Outcome: Change From Baseline in EuroQol Quality of Life Scale (EQ-5D) Summary Index at Endpoint
Description: The EQ-5D is a participant answered questionnaire scoring 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. EQ-5D health states, defined by the EQ-5D descriptive system, are converted into a single summary index by applying a formula that essentially attaches values (also called QOL weights or QOL utilities) to each of the levels in each dimension. EQ-5D Summary Index values range from -0.11 to 1.00 with positive change indicating improvement.
Time Frame: Baseline, Endpoint (last post-baseline visit up to Day 378)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Levodopa-Carbidopa Intestinal Gel (LCIG)
Number analyzed (Participants) | 313
units on a scale
  Baseline | 0.588 (0.195)
  Change from Baseline at Endpoint | 0.064 (0.203)
Statistical Analysis 1: Comparison: Levodopa-Carbidopa Intestinal Gel (LCIG); Test type: Superiority or Other; p < 0.001, t-test, 2 sided

31. Secondary Outcome: Change From Baseline in EuroQol Quality of Life Scale (EQ-5D) Visual Analogue Scale (VAS) at Endpoint
Description: The EQ-5D VAS records the participant's self-rated health on a scale from 0-100 where 100 is the 'best imaginable health state' and 0 is the 'worst imaginable health state'.
Time Frame: Baseline, Endpoint (last post-baseline visit up to Day 378)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Levodopa-Carbidopa Intestinal Gel (LCIG)
Number analyzed (Participants) | 313
units on a scale
  Baseline | 50.2 (21.0)
  Change from Baseline at Endpoint | 14.0 (24.8)
Statistical Analysis 1: Comparison: Levodopa-Carbidopa Intestinal Gel (LCIG); Test type: Superiority or Other; p < 0.001, t-test, 2 sided

32. Secondary Outcome: Change From Baseline in Zarit Burden Interview (ZBI) Total Score at Endpoint
Description: The ZBI is a 22-item questionnaire regarding the caregiver/subject relationship and evaluates the caregiver's health condition, psychological well-being, finances and social life. Each question is answered on a 5-point scale (0=never, 1=rarely, 2=sometimes, 3=quite frequently, and 4=nearly always). The caregiver burden is evaluated by the total score (Range 0 to 88) obtained from the sum of the answers to the 22 questions. Higher scores are associated with a higher level of burden for the caregiver.
Time Frame: Baseline, Endpoint (last post-baseline visit up to Day 378)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Levodopa-Carbidopa Intestinal Gel (LCIG)
Number analyzed (Participants) | 172
units on a scale
  Baseline | 27.1 (13.2)
  Change from Baseline at Endpoint | 0.2 (10.8)
Statistical Analysis 1: Comparison: Levodopa-Carbidopa Intestinal Gel (LCIG); Test type: Superiority or Other; p = 0.824, t-test, 2 sided

33. Primary Outcome: Number of Participants With Confirmed Cases of Melanoma
Description: A comprehensive assessment for the presence of melanoma was performed during the screening period and at early termination or end of study by a dermatologist experienced with the diagnosis of the condition. If a suspicious lesion was present, a biopsy was obtained for proper diagnosis.
Time Frame: Screening up to Day 378
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Levodopa-Carbidopa Intestinal Gel (LCIG)
Number analyzed (Participants) | 354
participants | 0

34. Primary Outcome: Number of Participants Taking at Least 1 Concomitant Medication During the Study
Description: Concomitant medications include those started on or after the first open-label LCIG infusion as well as medications started prior to the first open-label infusion but continued during the study.
Time Frame: Screening up to Day 378
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Levodopa-Carbidopa Intestinal Gel (LCIG)
Number analyzed (Participants) | 354
participants | 349

ADVERSE EVENTS:
Time Frame: From Screening to the end of study or early termination of treatment, including the removal of study device (up to 54 weeks), plus 30 days.
Description: Serious AEs and treatment-emergent AEs are presented. Treatment-emergent AEs were defined as AEs that began or worsened from date of the NJ device placement to the end of therapy (last dose of study drug or NJ/PEG-J removal, whichever is later) plus 30 days.
Arm/Group | Levodopa-Carbidopa Intestinal Gel (LCIG)
Serious Adverse Events (participants affected / at risk) | 108/354
Other Adverse Events (participants affected / at risk) | 278/354
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Levodopa-Carbidopa Intestinal Gel (LCIG) (N=354)
ANAEMIA (Blood and lymphatic system disorders) | 2
ANAEMIA VITAMIN B12 DEFICIENCY (Blood and lymphatic system disorders) | 1
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 1
ATRIOVENTRICULAR BLOCK SECOND DEGREE (Cardiac disorders) | 1
MYOCARDIAL INFARCTION (Cardiac disorders) | 1
SECONDARY ADRENOCORTICAL INSUFFICIENCY (Endocrine disorders) | 1
ANGLE CLOSURE GLAUCOMA (Eye disorders) | 1
CATARACT (Eye disorders) | 1
OPTIC ISCHAEMIC NEUROPATHY (Eye disorders) | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 10
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1
ACUTE ABDOMEN (Gastrointestinal disorders) | 2
BEZOAR (Gastrointestinal disorders) | 1
COLONIC POLYP (Gastrointestinal disorders) | 1
CONSTIPATION (Gastrointestinal disorders) | 2
DUODENAL PERFORATION (Gastrointestinal disorders) | 1
DYSPHAGIA (Gastrointestinal disorders) | 1
FAECALOMA (Gastrointestinal disorders) | 1
FLATULENCE (Gastrointestinal disorders) | 1
GASTRIC HYPOMOTILITY (Gastrointestinal disorders) | 1
GASTRITIS (Gastrointestinal disorders) | 1
HAEMORRHOIDAL HAEMORRHAGE (Gastrointestinal disorders) | 1
ILEUS PARALYTIC (Gastrointestinal disorders) | 1
INGUINAL HERNIA (Gastrointestinal disorders) | 1
INGUINAL HERNIA, OBSTRUCTIVE (Gastrointestinal disorders) | 1
INTESTINAL HAEMATOMA (Gastrointestinal disorders) | 1
INTESTINAL INFARCTION (Gastrointestinal disorders) | 1
INTESTINAL PERFORATION (Gastrointestinal disorders) | 1
INTESTINAL STENOSIS (Gastrointestinal disorders) | 1
LARGE INTESTINE PERFORATION (Gastrointestinal disorders) | 1
NAUSEA (Gastrointestinal disorders) | 2
PANCREATITIS (Gastrointestinal disorders) | 1
PERITONITIS (Gastrointestinal disorders) | 9
PNEUMATOSIS INTESTINALIS (Gastrointestinal disorders) | 1
PNEUMOPERITONEUM (Gastrointestinal disorders) | 8
SMALL INTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 2
VOMITING (Gastrointestinal disorders) | 1
ASTHENIA (General disorders) | 1
COMPLICATION OF DEVICE INSERTION (General disorders) | 21
DEATH (General disorders) | 2
DEVICE DISLOCATION (General disorders) | 5
DEVICE OCCLUSION (General disorders) | 3
IMPLANT SITE ULCER (General disorders) | 1
MEDICAL DEVICE COMPLICATION (General disorders) | 1
PAIN (General disorders) | 1
UNINTENTIONAL MEDICAL DEVICE REMOVAL BY PATIENT (General disorders) | 2
CHOLECYSTITIS (Hepatobiliary disorders) | 1
HEPATIC FAILURE (Hepatobiliary disorders) | 1
HEPATIC STEATOSIS (Hepatobiliary disorders) | 1
ABDOMINAL INFECTION (Infections and infestations) | 1
CLOSTRIDIUM DIFFICILE COLITIS (Infections and infestations) | 1
GASTROENTERITIS (Infections and infestations) | 1
GASTROENTERITIS VIRAL (Infections and infestations) | 1
LUNG ABSCESS (Infections and infestations) | 1
PERITONEAL ABSCESS (Infections and infestations) | 1
PNEUMONIA (Infections and infestations) | 7
POSTOPERATIVE WOUND INFECTION (Infections and infestations) | 3
PYELONEPHRITIS (Infections and infestations) | 2
PYELONEPHRITIS ACUTE (Infections and infestations) | 1
SEPSIS (Infections and infestations) | 1
SEPTIC SHOCK (Infections and infestations) | 1
URINARY TRACT INFECTION (Infections and infestations) | 1
UROSEPSIS (Infections and infestations) | 1
VIRAL DIARRHOEA (Infections and infestations) | 1
BRAIN CONTUSION (Injury, poisoning and procedural complications) | 1
CONTUSION (Injury, poisoning and procedural complications) | 2
FALL (Injury, poisoning and procedural complications) | 1
GASTROINTESTINAL STOMA COMPLICATION (Injury, poisoning and procedural complications) | 1
HIP FRACTURE (Injury, poisoning and procedural complications) | 6
LACERATION (Injury, poisoning and procedural complications) | 1
POST PROCEDURAL COMPLICATION (Injury, poisoning and procedural complications) | 2
POST PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 1
POSTOPERATIVE ILEUS (Injury, poisoning and procedural complications) | 1
RADIUS FRACTURE (Injury, poisoning and procedural complications) | 2
RIB FRACTURE (Injury, poisoning and procedural complications) | 1
STERNAL FRACTURE (Injury, poisoning and procedural complications) | 1
THORACIC VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 1
ULNA FRACTURE (Injury, poisoning and procedural complications) | 1
UPPER LIMB FRACTURE (Injury, poisoning and procedural complications) | 1
AMINO ACID LEVEL INCREASED (Investigations) | 1
BLOOD LACTIC ACID INCREASED (Investigations) | 1
WEIGHT DECREASED (Investigations) | 4
CACHEXIA (Metabolism and nutrition disorders) | 1
DECREASED APPETITE (Metabolism and nutrition disorders) | 1
FOLATE DEFICIENCY (Metabolism and nutrition disorders) | 1
HYPERHOMOCYSTEINAEMIA (Metabolism and nutrition disorders) | 1
HYPONATRAEMIA (Metabolism and nutrition disorders) | 1
MALNUTRITION (Metabolism and nutrition disorders) | 2
METABOLIC ACIDOSIS (Metabolism and nutrition disorders) | 1
VITAMIN B12 DEFICIENCY (Metabolism and nutrition disorders) | 1
VITAMIN B6 DEFICIENCY (Metabolism and nutrition disorders) | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 3
BURSITIS (Musculoskeletal and connective tissue disorders) | 1
RHABDOMYOLYSIS (Musculoskeletal and connective tissue disorders) | 1
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
BENIGN SALIVARY GLAND NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
COLON ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
RENAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
SQUAMOUS CELL CARCINOMA OF SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 1
DYSKINESIA (Nervous system disorders) | 1
GUILLAIN-BARRE SYNDROME (Nervous system disorders) | 2
HEADACHE (Nervous system disorders) | 1
HEPATIC ENCEPHALOPATHY (Nervous system disorders) | 1
HYPERKINESIA (Nervous system disorders) | 1
MONOPLEGIA (Nervous system disorders) | 1
MYELOPATHY (Nervous system disorders) | 1
NEUROPATHY PERIPHERAL (Nervous system disorders) | 1
ON AND OFF PHENOMENON (Nervous system disorders) | 2
PARKINSON'S DISEASE (Nervous system disorders) | 8
PARTIAL SEIZURES (Nervous system disorders) | 1
PERIPHERAL SENSORIMOTOR NEUROPATHY (Nervous system disorders) | 2
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 1
POLYNEUROPATHY (Nervous system disorders) | 9
SYNCOPE (Nervous system disorders) | 2
ACUTE PSYCHOSIS (Psychiatric disorders) | 1
AGITATION (Psychiatric disorders) | 1
ANXIETY (Psychiatric disorders) | 1
COMPLETED SUICIDE (Psychiatric disorders) | 2
DELUSION (Psychiatric disorders) | 1
DEPRESSION (Psychiatric disorders) | 4
HALLUCINATION (Psychiatric disorders) | 2
PSYCHOTIC DISORDER (Psychiatric disorders) | 2
STEREOTYPY (Psychiatric disorders) | 1
SUBSTANCE ABUSE (Psychiatric disorders) | 1
SUICIDE ATTEMPT (Psychiatric disorders) | 2
CALCULUS URETERIC (Renal and urinary disorders) | 2
NEPHROLITHIASIS (Renal and urinary disorders) | 1
RENAL FAILURE ACUTE (Renal and urinary disorders) | 1
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 1
PLEURISY (Respiratory, thoracic and mediastinal disorders) | 1
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 1
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 2
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 2
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1
EXCESSIVE GRANULATION TISSUE (Skin and subcutaneous tissue disorders) | 1
KNEE ARTHROPLASTY (Surgical and medical procedures) | 2
DEEP VEIN THROMBOSIS (Vascular disorders) | 1
HYPERTENSIVE CRISIS (Vascular disorders) | 1
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Levodopa-Carbidopa Intestinal Gel (LCIG) (N=354)
ABDOMINAL PAIN (Gastrointestinal disorders) | 92
CONSTIPATION (Gastrointestinal disorders) | 55
DIARRHOEA (Gastrointestinal disorders) | 27
DYSPEPSIA (Gastrointestinal disorders) | 24
NAUSEA (Gastrointestinal disorders) | 60
VOMITING (Gastrointestinal disorders) | 32
COMPLICATION OF DEVICE INSERTION (General disorders) | 102
POSTOPERATIVE WOUND INFECTION (Infections and infestations) | 47
URINARY TRACT INFECTION (Infections and infestations) | 37
FALL (Injury, poisoning and procedural complications) | 50
INCISION SITE ERYTHEMA (Injury, poisoning and procedural complications) | 43
INCISION SITE PAIN (Injury, poisoning and procedural complications) | 21
POST PROCEDURAL DISCHARGE (Injury, poisoning and procedural complications) | 26
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 67
PROCEDURAL SITE REACTION (Injury, poisoning and procedural complications) | 32
BLOOD HOMOCYSTEINE INCREASED (Investigations) | 20
VITAMIN B6 DECREASED (Investigations) | 20
WEIGHT DECREASED (Investigations) | 32
DECREASED APPETITE (Metabolism and nutrition disorders) | 18
BACK PAIN (Musculoskeletal and connective tissue disorders) | 23
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 19
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 19
DIZZINESS (Nervous system disorders) | 18
DYSKINESIA (Nervous system disorders) | 31
HEADACHE (Nervous system disorders) | 30
PARKINSON'S DISEASE (Nervous system disorders) | 25
ANXIETY (Psychiatric disorders) | 40
DEPRESSION (Psychiatric disorders) | 25
INSOMNIA (Psychiatric disorders) | 67
SLEEP ATTACKS (Psychiatric disorders) | 25
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 25
EXCESSIVE GRANULATION TISSUE (Skin and subcutaneous tissue disorders) | 51
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.